CLINICAL TRIAL: NCT01192724
Title: A Trial of Evaluating Additional Benefit of Cilostazol to Dual Antiplatelet Therapy in Patients With Long or Multi-vessel Coronary Artery Disease Underwent Biolimus-Eluting Stent Implantation
Brief Title: Additional Benefit of Cilostazol to Dual Antiplatelet Therapy After Biolimus-eluting Stent Implantation
Acronym: ABCD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Yoon Junghan, Junghan Yoon, M.D., Ph.D., Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABCD
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Coronary Artery Disease
Keywords: Antiplatelet; Coronary artery diseae; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Cilostazol; Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triple antiplatelet therapy (TAPT) group (Active Comparator): 3-month use of cilostazol in addition to dual antiplatelet agent
  Interventions: Drug: Cilostazol; Drug: Aspirin; Drug: Clopidogrel
- Dual antiplatelet therapy (DAPT) group (Active Comparator): Aspirin and clopidogrel (dual antiplatelet therapy, DAPT) for 1 year
  Interventions: Drug: Aspirin; Drug: Clopidogrel

INTERVENTIONS:
Drug: Cilostazol — 100 mg BID, for 3 months
  Other Names: pletaal
  Arms: Triple antiplatelet therapy (TAPT) group
Drug: Aspirin — Aspirin 100 mg QD, for 1 year
  Other Names: Aspirin protect; Astrix; Baby rhonal
Drug: Clopidogrel — Clopidogrel 75 mg QD, for 1 year
  Other Names: Plavix; Plavitor; Platless

SUMMARY:
Because there is limited data about long-term efficacy and safety about short-term use of cilostazol adding to dual antiplatelet therapy in patients with long or multivessel coronary artery disease after 2nd generation DES implantation, especially in biodegradable polymer stent, the investigators will evaluate whether a 3-month use of cilostazol in addition to dual antiplatelet therapy effectively reduces clinical adverse outcome at 1 year in subject with long or multivessel coronary artery disease after biolimus-eluting stent implantation.

DETAILED DESCRIPTION:
Previous randomized trials have shown the efficacy of drug-eluting stent (DES) such as sirolimus-eluting stent (CYPHERTM, Cordis, Warren, NJ, USA), paclitaxel-eluting stent (TAXUSTM, BostonScientific, Natick, MA, USA), and zotarolimus-eluting stent (Endeavor,Medtronic,Minneapolis, MN, USA) over bare metal stents (BMS) in reducing neointimal hyperplasia, late luminal loss, and angiographic restenosis leading to decreased target lesion revascularization.1-4 In addition, Among patients with off-label indications, the use of DESs reduced a rate of repeat revascularization without increasing the risk of death or myocardial infarction, as compared with bare-metal stents.5 But, compared with on-label use, off-label use of DESs is associated with a higher rate of adverse outcomes such as death, myocardial infarction and target vessel revascularization. Furthermore, stent thrombosis (ST) occurred predominantly in patients who underwent off-label DES implantation.6 It is known that the risk of adverse cardiac events and ST after DES implantation is related to stent length.7 Cilostazol is a potent phosphodiesterase III inhibitor preventing the hydrolysis of cAMP in platelets and vascular smooth muscle cell. The novel mechanism of action of cilostazol reduces the number of circulating, partially activated, or preconditioned platelets, by reducing the surface expression of adhesive molecules in endothelial cells interacting with circulating platelets. The agent also directly inhibits platelet aggregation induced by a variety of stimuli, including arachidonic acid, ADP, collagen, thrombin, and high shear stress.8 In current guidelines, a 12-month duration of dual antiplatelet therapy with aspirin and clopidogrel is recommended after DES implantation.9 But, recent meta-analyses showed a potential benefit of cilostazol in addition to dual antiplatelet therapy in reducing angiographic restenosis and improved clinical outcomes after BMS or DES implantation.10, 11 Actually, additional cilostazol to dual antiplatelet therapy showed reduced restenosis and late loss in patients with long coronary lesion and diabetes with multivessel coronary artery disease and it also showed beneficial effect on stent thrombosis after DES implantation.12-14 Although most studies showed no difference in bleeding according to additional cilostazol to dual antiplatelet therapy, the rate of early cessation of cilostazol due to adverse effect including headache, palpitation, skin rash and hepatic dysfunction was about 15%.12-14 Because of relatively higher side effect rate and no definitive duration of addition cilostazol use, we expect that cilostazol with short duration can be easily accepted to patient. Although almost studies about cilostazol after stent implantation used a 6- month duration of cilostazol, one study showed that use of cilostazol for 3 months after percutaneous transluminal coronary balloon angioplasty reduced restenosis and revascularization, as compared with use of aspirin.15 So, we expect a 3-month use of additional cilostazol to dual antiplatelet therapy can reduce the adverse outcome and ST after stent implantation without increasing early cessation of cilostazol.

The BioMatrixTM stent system (Biosensors Interventional Technologies Pte., Ltd, Singapore) consist of a stainless steel, quadrature-link design, balloon expandable S-StentTM, and a polylactic acid (PLA) polymer and BiolimusA9® coating mounted on a low-profile delivery catheter.16, 17 It is expected that abluminal biodegradable coating of BioMatrixTM stent can lead to more targeted drug release, reduced systemic exposure and early BMS-like endothelial coverage.18 The first-in-man, randomized controlled SEALTH I trial demonstrate higher efficacy of BioMatrixTM stent by showing lower late lumen loss and in-stent restenosis as compared with BMS, S-stent at 6-month follow-up.19 In LEADERS trial, BioMatrixTM stent showed similar efficacy and safety as compared with sirolimus-eluting stent in patients with chronic stable coronary artery disease and acute coronary syndromes.20 But significantly lower uncovered and malapposed struts was detected by optical coherence tomography study.21 This means more complete coverage of struts and we can expect lower late ST after BioMatrixTM stent implantation.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years.
* Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving the BioMatrix® and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
* Subject must have significant coronary artery stenosis (>70% by visual estimate).
* Subject must have evidence of myocardial ischemia (e.g., stable, unstable angina, recent infarction, acute myocardial infarction, silent ischemia, positive functional study or a reversible changes in the ECG consistent with ischemia).
* Target lesion(s) located in a native coronary artery with visually estimated diameter of ≥ 2.0 and ≤ 4.24 mm
* Target lesion(s) amenable for PCI
* Lesion(s) must have at least 1 of these 2 angiographic features to be eligible
* Lesion(s) need(s) stent length ≥ 28mm (multiple stents whether are overlapped or not are allowed. No limitation of stent length)
* Multivessel coronary artery disease that need ≥2 stents regardless of stent length
* Significant (>70%) lesions in at least two major epicardial vessels (≥ 2.0mm in diameter)
* Lesion(s) of chronic total occlusion or bifurcation which need ≥ 2 stents can be eligible

Exclusion criteria:

* The subject has a known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel, biolimus A9, stainless steel, cobalt chromium, contrast media*. (*Subjects with documented sensitivity to contrast media, which can be effectively premedicated with steroid and diphenhydramine may be enrolled. However, those with true anaphylaxis to prior contrast media should not be enrolled.)
* Systemic (intravenous) biolimus A9 use within 12 months.
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
* History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions.
* Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months.
* Current known current platelet count <100,000 cells/mm3 or Hgb <10 g/dL.
* An elective surgical procedure is planned that would necessitate interruption of thienopyridines during the first 12 months post enrollment
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Subjects who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
* Subjects who have received DES implantation in the any coronary artery prior to enrollment
* Subjects with heart failure, NYHA class III or IV or those with cardiogenic shock. (The degree of left ventricular ejection fraction is not considered as an index of exclusion)
* Creatinine level > 3.0mg/dL or dependence on dialysis.
* Severe hepatic dysfunction AST or ALT > 3 times upper normal reference values) except MI-induced elevation
* Subjects who need antagonist of vitamin K due during study
* Isolated left main disease (lesion(s) at proximal LAD or LCX lesion that need to cross the left main can be enrolled)
* Target lesion(s) with ISR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Device-oriented composite | One year
  Device-oriented composite was defined as a composite of cardiac death, MI (not clearly attributable to a non-target vessel), and clinically indicated target lesion revascularization (TLR).

SECONDARY OUTCOMES:
Patient-oriented composite | One year
  Patient-oriented composite was defined as a composite of all-cause mortality, any MI (includes non-target vessel territory), and any repeat revascularization (includes all target and non-target vessel).
Each component of device- and patient-oriented composite | One year
  All-cause mortality, cardiac death, any myocardial infarction (MI), MI (not clearly attributable to a non-target vessel), clinically indicated target lesion revascularization (TLR), and any repeat revascularization (includes all target and non-target vessel)
Academic Research Consortium (ARC) defined stent thrombosis | One year
  definite, probable, and possible stent thrombosis / acute, subacute, and late stent thrombosis
Safety assessments | One year
  Safety assessments will be performed for bleeding complication according to Thrombolysis In Myocardial Infarction (TIMI) criteria, medication compliance, side effect of drug, and heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: Junghan Yoon, M.D., Ph.D., Principal Investigator — Wonju College of Medicine, Yonsei University
Locations (1):
- Wonju Christian Hospital, Wŏnju, Gangwon-do, South Korea

REFERENCES:
- [Result] Youn YJ, Lee JW, Ahn SG, Lee SH, Choi H, Yu CW, Hong YJ, Kwon HM, Hong MK, Jang Y, Yoon J. Multicenter randomized trial of 3-month cilostazol use in addition to dual antiplatelet therapy after biolimus-eluting stent implantation for long or multivessel coronary artery disease. Am Heart J. 2014 Feb;167(2):241-248.e1. doi: 10.1016/j.ahj.2013.08.028. Epub 2013 Oct 22. PMID 24439986